CLINICAL TRIAL: NCT05808725
Title: Relative Bioavailability Study of Amlodipine Powder for Oral Solution, 5 mg (Base) Under Fasting and Fed Conditions
Brief Title: Amlodipine Freeze-Dried Powder for Oral Solution 5 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brillian Pharma Inc. (Industry)
Collaborators: Accutest Research Laboratories (I) Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ARL-22-073
Record Dates: First submitted 2023-03-07; First posted 2023-04-11 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Hypertension; Coronary Artery Disease
MeSH Terms: conditions — Hypertension; Coronary Artery Disease | interventions — Solutions; Amlodipine

STUDY DESIGN:
Intervention Model Description: A Randomized, Open Label, Balanced, Three Treatment, Three period, Three Sequence, Single Dose, Crossover design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- T1 Fasting (Experimental): Giving test product under fasting condition
  Interventions: Drug: Amlodipine Freeze-Dried Powder for Oral Solution 5 mg
- T2 Fed (Experimental): Giving test product under fed condition
  Interventions: Drug: Amlodipine Freeze-Dried Powder for Oral Solution 5 mg
- R Fasting (Active Comparator): Giving reference product under fasting condition
  Interventions: Drug: Norvasc 5 mg tablets of Pfizer Labs

INTERVENTIONS:
Drug: Amlodipine Freeze-Dried Powder for Oral Solution 5 mg — Amlodipine Oral Solution 5 mg is given to T1 Fasting and T2 Fed
  Other Names: Amlodipine Oral Solution 5 mg
  Arms: T1 Fasting; T2 Fed
Drug: Norvasc 5 mg tablets of Pfizer Labs — Norvasc 5 mg is given to R Fasting
  Other Names: Amlodipine Besylate 5 mg
  Arms: R Fasting

SUMMARY:
The goal of this clinical study is to assess the relative bioavailability of Amlodipine for Oral Solution 5 mg of Brillian Pharma Inc. under fasting and fed conditions versus reference product Norvasc 5 mg tablets of Pfizer Labs under fasting in normal, healthy, adult, male,

Primary Objective:

1. To compare the relative bioavailability.
2. To assess the food effect in Test product (T1) (Fast) vs Test product (T2) (Fed) Amlodipine Oral Solution 5 mg of Brillian Pharma Inc.

Secondary Objective:

To monitor the safety and tolerability of a single oral dose of investigational medicinal products (IMPs).

DETAILED DESCRIPTION:
A total of 24 healthy, adult, male and female human volunteers will be enrolled.

Excluding the screening period, the duration of the clinical phase will be approximately 50 days including a washout period of at least 21 days for each study period.

This study is being conducted in healthy, adult, human subjects under fasting and fed conditions as per USFDA and NMPA guidelines. The present study will be conducted to assess the relative bioavailability of the test product versus the reference product under fasting conditions. The study also assesses the effect of food on the bioavailability of Amlodipine FD-POS 5 mg (Powder in a Unit-dose container) product.

ELIGIBILITY:
Inclusion Criteria:

* Adult, Healthy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Cmax | 1, 2, 3, 4, 5,6, 7, 8, 9, 10, 12, 14, 16, 20, 24, 48, 60, 72, 96, 120, 144 hours post dose
  Maximum observed drug concentration during the study
AUC0-t | 50 days
  Area under the plasma concentration-time curve measured to the last quantifiable concentration, using the linear trapezoidal rule.
AUC0-inf | 1, 2, 3, 4, 5,6, 7, 8, 9, 10, 12, 14, 16, 20, 24, 48, 60, 72, 96, 120, 144 hours post dose
  AUC0-t plus additional area extrapolated to infinity, calculated using the formula AUC0-t + Ct/Kel , where Ct is the last measurable drug concentration and Kel is the elimination rate constant.

SECONDARY OUTCOMES:
Tmax | 6 days
  Time to observe maximum drug concentration. If the maximum value occurs at more than 1 time point, Tmax is defined as the first time point with this value.
AUC0-t/AUC0-inf | 1, 2, 3, 4, 5,6, 7, 8, 9, 10, 12, 14, 16, 20, 24, 48, 60, 72, 96, 120, 144 hours post dose
  Ratio of AUC0-t and AUC0-inf
Residual Area | 1, 2, 3, 4, 5,6, 7, 8, 9, 10, 12, 14, 16, 20, 24, 48, 60, 72, 96, 120, 144 hours post dose
  Extrapolated area (AUC0-inf - AUC0-t)/ AUC0-inf
Kel | 6 days
  Apparent first - order terminal elimination rate constant calculated from a semi-log plot of the plasma concentration versus time curve, using the method of least square regression.
t1/2 | 6 days
  Terminal half-life as determined by quotient 0.693/Kel

CONTACTS AND LOCATIONS:
Overall Officials: Pratikkumar Dilipbhai Asari, M.D., Principal Investigator — Accutest Research Laboratories (I) Pvt. Ltd.
Locations (1):
- Accutest Research Laboratories (I) Pvt. Ltd., Vadodara, Gujarat, India

IPD SHARING:
Plan to Share IPD: No